CLINICAL TRIAL: NCT02270060
Title: The Effects of a Single Music Therapy Session on the Pain of Adult Patients With Sickle Cell Disease: A Mixed Methods Study
Brief Title: Music Therapy in Sickle Cell Pain Mixed Methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Music Therapist, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-14-11
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Sickle Cell Disease
Keywords: Music Therapy; Sickle Cell Disease; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Music Therapy Group (Experimental): Patient receives a single 20-minute music therapy session with a music therapist. Patient will interact with specially composed music tailored to the patient's preferences using an iPad.
  Interventions: Other: Music Therapy
- Music Listening Group (Active Comparator): Patient listens to his/her preferred music on an iPod touch for 20 minutes without the presence of a music therapist.
  Interventions: Other: Music Listening
- Control Group (No Intervention): Patient receives standard care and waits in treatment room/bay for twenty minutes.

INTERVENTIONS:
Other: Music Therapy — Patient receives a single 20-minute music therapy session with a music therapist. Patient will interact with specially composed music tailored to the patient's preferences using an iPad.
  Arms: Music Therapy Group
Other: Music Listening — Patient listens to his/her preferred music on an iPod touch for 20 minutes without the presence of a music therapist.
  Arms: Music Listening Group

SUMMARY:
The purpose of this research study is to:

1. Investigate the effects of a single 20-minute music therapy intervention with a music therapist on the pain intensity, pain relief, and mood of adult patients with sickle cell disease as compared to:

   1. Adult patients with SCD who listen to their preferred music for 20 minutes without the presence of a music therapist (music listening group)
   2. Adult patients with SCD who receive standard care alone (control group)
2. Determine the feasibility (delivery, acceptability, and usefulness) of the music therapy intervention for pain management

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a diagnosis of sickle cell disease (HbSS, HbSC, HbSbeta+thal, or HbSbeta0thal)
* 18 years or older
* Able to speak and understand English

Exclusion Criteria:

* Patients who have significant hearing impairments and/or significant visual impairments that have not been corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel N Rodgers-Melnick, MT-BC, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following verbal consent on the day of an ACC visit, an RN escorted the participant into the ACC to receive standard care that included vital signs, a lab draw, assessment by a nurse practitioner, and scheduled analgesics. The assigned study condition occurred one hour after participants' first dose of analgesics.
Period: Overall Study
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Therapy Group | Music Listening Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.85 (9.49) | 33.25 (11.23) | 30.60 (7.44) | 31.57 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 35
  Male | 8 | 9 | 8 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 20 | 20 | 60
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Type of Sickle Cell Disease [Count of Participants; unit: Participants]
  HbSS | 10 | 15 | 12 | 37
  HbSC | 6 | 4 | 5 | 15
  HbSbeta+ Thalassemia | 3 | 0 | 3 | 6
  HbSbeta0 Thalassemia | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change (Post - Pre) From Baseline in Visual Analog Scale of Pain Intensity (VASPI) of Memorial Pain Assessment Card
Description: Visual analog scale of pain intensity. The minimum score is 0. The maximum score is 10. Higher scores represent worse pain intensity.
Time Frame: Baseline and at end of 20-minute intervention, up to 120 minutes following randomization
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | -1.92 (1.88) | -1.92 (2.50) | -1.19 (1.69)

2. Secondary Outcome: Change (Post - Pre) From Baseline in Visual Analog Scale of Pain Relief (VASPR) of Memorial Pain Assessment Card
Description: Visual analog scale of Pain Relief. The minimum score is 0. The maximum score is 10. Higher scores represent greater pain relief.
Time Frame: Baseline and at end of 20-minute intervention, up to 120 minutes following randomization
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 2.05 (2.33) | .86 (4.01) | .45 (1.97)

3. Secondary Outcome: Change (Post- Pre) From Baseline in Visual Analog Scale of Mood (VASMOOD) of Memorial Pain Assessment Card
Description: Visual analog scale of mood. The minimum score is 0. The maximum score is 10. Higher scores represent better mood.
Time Frame: Baseline and at end of 20-minute intervention, up to 120 minutes following randomization
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 2.33 (2.10) | .96 (2.38) | .74 (1.98)

4. Secondary Outcome: Change (Post - Pre) From Baseline in Tursky Scale of Memorial Pain Assessment Card
Description: Pain adjectives scale. The minimum score is 1. The maximum score is 7. Higher scores represent worse pain.
Time Frame: Baseline and at end of 20-minute intervention, up to 120 minutes following randomization
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | -0.80 (1.20) | -0.35 (2.23) | -0.50 (1.00)

5. Secondary Outcome: Length of Stay in Minutes
Description: Length of stay (in minutes) in acute care clinic
Time Frame: From time of admission into acute care clinic to time of discharge, up to 8 hours.
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
minutes | 272.95 (72.84) | 286.80 (116.74) | 287.45 (119.75)

6. Secondary Outcome: Amount of Hydromorphone
Description: Amount of Hydromorphone received in acute care clinic following intervention
Time Frame: From time of admission into acute care clinic to time of discharge, up to 8 hours.
Population: All participants who participated in the music therapy intervention and received hydromorphone.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 19 | 18 | 18
milligrams | 10.30 (7.84) | 8.10 (6.70) | 10.00 (8.25)

7. Secondary Outcome: Change (Post - Pre) From Baseline in Numeric Pain Rating (NPR)
Description: Numeric pain rating between 0-10 before and after admission to acute care clinic. The minimum score is 0. The maximum score is 10. Higher scores represent worse pain.
Time Frame: From time of admission into acute care clinic to time of discharge, up to 8 hours.
Population: All participants who participated in the music therapy intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | -2.70 (1.63) | -2.95 (1.68) | -3.10 (1.97)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 20 month study period. For each participant, adverse event data was collected between baseline measurement of clinical outcomes and the end of each participant's participation in the study in the acute care clinic. This duration varied between 2 and 6 hours for each participant depending on his/her length of stay.
Arm/Group | Music Therapy Group | Music Listening Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Small sample size and potential risk of bias, due to some participants having previous clinical relationships with the investigators prior to study initiation. We were unable to blind participants to their study condition assignments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes